CLINICAL TRIAL: NCT04621695
Title: Comparison of Rubber Band Ligation and Haemorrhoidectomy in Patients With Symptomatic Haemorrhoids Grade III: a Multicentre, Randomized Controlled Trial and Cost-utility Analysis.
Brief Title: Comparison of Rubber Band Ligation and Haemorrhoidectomy in Patients With Symptomatic Haemorrhoids Grade III
Acronym: HollAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Proctos Kliniek (Other)
Responsible Party: Principal Investigator, dr. IJM Han-Geurts, Principal investigator, Proctos Kliniek
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL69227.018.19
Record Dates: First submitted 2020-10-23; First posted 2020-11-09 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Hemorrhoids; Hemorrhoids, Internal; PROM; Rectal Diseases
Keywords: Hemorrhoids; Hemorrhoidal disease; Rubber band ligation; Hemorrhoidectomy; PROM
MeSH Terms: conditions — Hemorrhoids; Rectal Diseases | interventions — Hemorrhoidectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rubber band ligation (Other): Rubber band ligation is performed by a suction device that allows a rubber band to be applied at the base of the haemorrhoid via a proctoscope. Maximal suction force used is 40 mmHg. A maximum of 3-4 bands are used per session. This rubber band constricts the blood supply causing it to become ischaemic before being sloughed approximately 1-2 weeks later. The resultant fibrosis reduces any element of haemorrhoidal prolapse that may have been present. No sedation is required for this day-care procedure. Patients are asked to administer an enema 2 hours prior to the procedure.
  Interventions: Procedure: RBL
- Hemorrhoidectomy (Other): There are two main excisional procedures currently carried out: open (Milligan and Morgan) and closed (Ferguson). Both have the intention of excising the haemorrhoidal cushions. The procedure is performed under either general or spinal anaesthesia in a day-care setting.
  Patients were asked to administer an enema 2 hours prior to the procedure.
  Interventions: Procedure: Hemorrhoidectomy

INTERVENTIONS:
Procedure: RBL — Both arms are standard care procedures in the Netherlands
  Arms: Rubber band ligation
Procedure: Hemorrhoidectomy — Both arms are standard care procedures in the Netherlands
  Arms: Hemorrhoidectomy

SUMMARY:
Rationale: Haemorrhoidal disease is one of the most common anorectal disorders which affects nearly half of the general population1. Given the current numerous modalities the obvious question which needs to be answered is which treatment is the best. An interesting conclusion from a recent systematic review regarding operative procedures for haemorrhoidal disease is that all procedures have their own advantages and disadvantages. There is a need for evaluating treatment from the patient's point of view and transparency in surgical and non-surgical treatment outcome. So far there is no sufficiently large trial that meets that demand.

Objective: To establish the best treatment of patients with symptomatic haemorrhoids grade III: haemorrhoidectomy versus rubber band ligation (RBL). Patient bound effectiveness, clinical effectiveness and cost-utility of both treatments is compared; primary outcome is quality of life at 24 months measured with the EQ-5D-5L with Dutch rating and recurrence at one year post procedure. The assumption is that treatment with rubber band ligation is equally effective in comparison with haemorrhoidectomy in terms of quality of life.

Study design:Multicentre randomized controlled non-inferiority trial with cost-utility analysis. Two treatment protocols are compared: haemorrhoidectomy and rubber band ligation.

Study population: Patients aged ≥ 18 years with symptomatic haemorrhoids gr III. Patients are recruited in multiple clinics during 18-24 months.

Intervention: Participants are allocated to either rubber band ligation or haemorrhoidectomy.

Main study parameters/endpoints: Primary outcome measure is quality of life at 24 months measured with the EQ-5D-5L with Dutch rating and recurrence at one year post procedure. Secondary outcomes are: complaint reduction with proctology specific patient-related outcome measure (HSS, PROM, PROMHISS), vaizey score, resumption of work, pain (VAS), complications and recurrence at two years.

ELIGIBILITY:
Inclusion Criteria:

* Haemorrhoids grade III (Goligher classification)
* Age 18 years and older
* Sufficient understanding of the Dutch written language (reading and writing)

Exclusion Criteria:

* Previous rectal or anal surgery with the exception of rubber band ligation
* Previous surgery for haemorrhoids (at any time)
* More than one injection treatment for haemorrhoids in the past 3 years
* More than one rubber band ligation procedure in the past 3 years
* Previous rectal radiation
* Pre-existing sphincter injury
* Inflammatory bowel disease
* Medically unfit for surgery or for completion of the trial (ASA>III)
* Pregnancy
* Hyper-coagulability disorders
* Patients previously randomised to this trial
* Not able or willing to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-11-25 (Estimated); Study Completion 2023-11-25 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | 24 months
  The EQ-5D-5L is a generic Health Related Quality of Life (HRQoL) measure, which is broadly used in economic evaluation. The instrument examines a patient's HRQoL on the day of the interview. It consists of the EQ-5D-5L descriptive system and the EQ-Visual Analogue Scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses to the 5 items result in a patient's health state that can be transformed into an index score representing health-related quality of life, ranging between 0 (death) and 1 (full health). These index scores are combined with length of life to calculate the QALY. The EQ-VAS records the patient's self-rated health with endpoints labelled 'the best health you can imagine' at the top and 'the worst health you can imagine' at the bottom.
Recurrence | at 12 months
  Patient self reported assessment with a dichotomous question: "At the moment, do you feel your symptoms from your haemorrhoids are: (1) cured or improved compared with before treatment; or (2) unchanged or worse compared with before treatment?" Any patient who answers '1' but has required further treatment since the initial procedure will be reclassified as '2', identified via hospital records, their consultant and patient questioning
In-hospital direct costs | this will be asked at 6 weeks, 6, 12 and 24 months
  with EQ-5D-5L and cost incremental analysis (iMCQ and iPCQ): The impact of disease on the ability of a person to perform work should be part of an economic evaluation when a societal perspective is applied. iMTA is highly experienced in methods for measuring and valuing productivity losses.The Productivity Costs Questionnaire (iPCQ) may be combined with the iMTA Medical Consumption Questionnaire (iMCQ), a generic instrument for measuring medical costs. The iMCQ includes questions related to frequently occurring contacts with health care providers and can be complemented with extra questions that are relevant for specific study populations.
In-hospital indirect costs | this will be asked at 6 weeks, 6, 12 and 24 months
  with EQ-5D-5L and cost incremental analysis (iMCQ and iPCQ): The impact of disease on the ability of a person to perform work should be part of an economic evaluation when a societal perspective is applied. iMTA is highly experienced in methods for measuring and valuing productivity losses.The Productivity Costs Questionnaire (iPCQ) may be combined with the iMTA Medical Consumption Questionnaire (iMCQ), a generic instrument for measuring medical costs. The iMCQ includes questions related to frequently occurring contacts with health care providers and can be complemented with extra questions that are relevant for specific study populations.
Out-of-hospital postoperative costs | this will be asked at 6 weeks, 6, 12 and 24 months
  with EQ-5D-5L and cost incremental analysis (iMCQ and iPCQ): The impact of disease on the ability of a person to perform work should be part of an economic evaluation when a societal perspective is applied. iMTA is highly experienced in methods for measuring and valuing productivity losses.The Productivity Costs Questionnaire (iPCQ) may be combined with the iMTA Medical Consumption Questionnaire (iMCQ), a generic instrument for measuring medical costs. The iMCQ includes questions related to frequently occurring contacts with health care providers and can be complemented with extra questions that are relevant for specific study populations.

SECONDARY OUTCOMES:
Health related quality of life | 12 months
  The EQ-5D-5L is a generic Health Related Quality of Life (HRQoL) measure, which is broadly used in economic evaluation. The instrument examines a patient's HRQoL on the day of the interview. It consists of the EQ-5D-5L descriptive system and the EQ-Visual Analogue Scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses to the 5 items result in a patient's health state that can be transformed into an index score representing health-related quality of life, ranging between 0 (death) and 1 (full health). These index scores are combined with length of life to calculate the QALY. The EQ-VAS records the patient's self-rated health with endpoints labelled 'the best health you can imagine' at the top and 'the worst health you can imagine' at the bottom.
Patient reported outcome measures concerning symptoms in daily life; Vaizey score | 12 months
  Vaizey faecal continence score consists of 7 questions with a maximum of score of 24. The higher the score, the higher the worse the outcome.
Patient reported outcome measures concerning symptoms in daily life; proctoPROM | 12 months
  The proctoPROM is a validated questionnaire consisting of five questions concerning patients well-being, wich are each scored on a numeric rating scale from 0 to 10. Regarding impact of symptoms, 0 correlates with 'no impact at all' and 10 with 'highly impacted on daily life'. Than the mean of the 5 question is taken.
Patient reported outcome measures concerning symptoms in daily life; PROM-HISS | 12 months
  Patient-Reported Outcome Measure-Haemorrhoidal Impact and Satisfaction Score which are each scored on a numeric rating scale from 0 to 10. Regarding impact of symptoms, 0 correlates with 'no impact at all' and 10 with 'highly impacted on daily life'. For patient satisfaction with treatment, this ranges between 0 'not satisfied' and 10 'very satisfied'.
Patient reported outcome measures concerning symptoms in daily life; HHS | 12 months
  Hemorrhoid severity score consists of five questions concerning the frequency of symptoms of hemorrhoids. The higher the score the more frequent the symptoms occur.
Patient reported outcome measures concerning symptoms in daily life, VAS pain score | this will be asked 1 day post procedure, 1 week and 6 weeks post procedure.
  The pain visual analogue scale has a numeric rating scale from 0 to 10 with 0 being 'no pain' and 10 'worse pain you ever felt'.
Return to work | this will be asked at 1 week and 6 weeks post procedure.
  Number of days patients are able to return to work
Need for further treatment | 12 months
Complications | 12 months
  Adverse events as: peroperative bleeding, postoperative bleeding, urinary retention requiring catheterisation, pelvic sepsis, anal fissure, anal fistula, wound discharge, residual anal skintages, anal stenosis, fecal incontinence, death

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Han-Geurts, MD PhD, Principal Investigator — Proctos Kliniek; Willem Bemelman, Prof., Study Chair — Amsterdam University Medical Center, location AMC
Locations (9):
- Netherlands (9):
  - Flevoziekenhuis, Almere Stad
  - Meander MC, Amersfoort
  - OLVG, Amsterdam
  - University Medical Center location AMC, Amsterdam
  - IJsselland ziekenhuis, Capelle aan den IJssel
  - Groene Hart ziekenhuis, Gouda
  - MUMC+, Maastricht
  - Centraal Militair Hospitaal, Utrecht
  - Diakonessenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
(Several versions of) processed data, documentation of the research process, including deindentified participant data, raw data, syntaxes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months embargo due to publishing.
Access Criteria: There will be access restrictions to my data collection. A request must be made at Data Access Committee (DAC).

REFERENCES:
- [Derived] van Oostendorp JY, Dekker L, van Dieren S, Veldkamp R, Bemelman WA, Han-Geurts IJM; HOLLAND study group. Cost-Effectiveness of Rubber Band Ligation Versus Hemorrhoidectomy for the Treatment of Grade III Hemorrhoids: Analysis Using Evidence From the HOLLAND Randomized Controlled Trial. Dis Colon Rectum. 2025 Sep 1;68(9):1100-1111. doi: 10.1097/DCR.0000000000003832. Epub 2025 Jun 10. PMID 40492557
- [Derived] van Oostendorp JY, Dekker L, van Dieren S, Veldkamp R, Bemelman WA, Han-Geurts IJM; HollAND Study Group. Comparison of Rubber Band Ligation and Hemorrhoidectomy in Patients With Symptomatic Hemorrhoids Grade III: A Multicenter, Open-Label, Randomized Controlled Noninferiority Trial. Dis Colon Rectum. 2025 May 1;68(5):572-583. doi: 10.1097/DCR.0000000000003679. Epub 2025 Feb 14. PMID 39952268
- See also: Study website — http://zorgevaluatienederland.nl/holland